CLINICAL TRIAL: NCT02746263
Title: A Randomized, Double-Blind, Double-Dummy, Active-Controlled, Repeated Dose, Multicenter Study to Compare Intravenous and Oral Acetaminophen for the Treatment of Acute Moderate to Severe Pain in Combination With Patient-Controlled Analgesia With Morphine in Adults Following Elective Total Knee Arthroplasty
Brief Title: Multicenter Study to Compare Intravenous and Oral Acetaminophen for the Treatment of Acute Moderate to Severe Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision because enrollment was slower than expected
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MNK14504054
Record Dates: First submitted 2016-03-18; First posted 2016-04-21 (Estimated); Results first posted 2019-11-06 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2016-11

CONDITIONS: Acute Pain, Postoperative
Keywords: Elective total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV acetaminophen/Morphine (Experimental): IV acetaminophen 1000 mg every 6 hours over 18 hours
  Interventions: Drug: IV acetaminophen; Drug: Morphine
- Oral acetaminophen/Morphine (Active Comparator): Oral acetaminophen two 500 mg tablets every 6 hours over 18 hours
  Interventions: Drug: Oral acetaminophen; Drug: Morphine

INTERVENTIONS:
Drug: IV acetaminophen
  Other Names: Ofirmev
  Arms: IV acetaminophen/Morphine
Drug: Oral acetaminophen
  Other Names: Acetaminophen (APAP)
  Arms: Oral acetaminophen/Morphine
Drug: Morphine — Patient controlled analgesia

SUMMARY:
The purpose of this study is to compare intravenous (IV) and oral acetaminophen for the treatment of acute moderate to severe pain in combination with standard patient-controlled analgesia (PCA) in adult subjects following total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be adequately informed and understand the nature and risks of the study and must be able to provide a signature and date on the informed consent form.
2. Subject must be male or females, between 50 and 90 years of age (inclusive) at Screening.
3. Subject must have a weight range of 50 to 120 kg.
4. Subject must be in a American Society of Anesthesiologists risk class of I, II, or III.
5. Subject must have successfully completed an unilateral uncomplicated total knee replacement surgery, able to take oral medication, and report having moderate to severe acute pain as determined by a pain score ≥ 5 from the 11-point Numeric Pain Rating Scale (NPRS) scale during the period of 3 to 6 hours postsurgery.
6. Female subjects of child-bearing potential must have a negative serum pregnancy test at the Screening and day-of-surgery.
7. Subjects must be able to communicate effectively with study personnel.
8. Subject must be able and willing to follow all protocol requirements, including operating a PCA device, and study restrictions.

Exclusion Criteria:

1. Subject is from a vulnerable population, as defined by the Code of Federal Regulations Title 45, Part 46, 1. Section 46.111(b), including but not limited to employees (temporary, part-time, full time, etc.) or a family member of the research staff conducting the study, or of the sponsor, or of the clinical research organization, or of the Institutional Review Board.
2. Subject has an oxygen saturation of less than 95% while awake on room air.
3. Subject has a positive test result for human immunodeficiency virus, hepatitis B (surface antigen), or hepatitis C virus antibody at Screening.
4. Subject has used an average of 30 mg oral morphine equivalents or greater, 1 to 2 weeks prior to the day of surgery. Subjects who, in the investigator's opinion are developing opioid tolerance will be excluded.
5. Subject has a history of any drug allergy, hypersensitivity, or intolerance to acetaminophen or morphine or to any of the excipients in the IV or oral formulations used.
6. Subject has intra- or postoperative complications, which in the view of the investigator, makes the subject unsuitable for the participation of the study.
7. Subject has received neuraxial (spinal or epidural) opioid injected perioperatively.
8. Subject has received a local anesthetic, regional, or wound injection or continuous infusion by any route.
9. Subject has impaired liver function (eg, aspartate aminotransferase, alanine aminotransferase, or bilirubin greater than or equal to 3.0 times the upper limit of normal), active hepatic disease, evidence of clinically significant liver disease, or other condition (eg, alcoholism, cirrhosis, or hepatitis) that suggests the potential for an increased susceptibility to hepatic toxicity with study drug exposure.
10. Subject has renal dysfunction or is at risk for renal failure due to volume depletion.
11. Subject has donated or had significant loss of whole blood (480 mL or more) within 30 days, or plasma within 14 days prior to dosing.
12. Subject has had any major surgery within 3 months prior to day-of-surgery.
13. Subject has a history of acute illness within 14 days prior to day-of-surgery.
14. Subject has participated in another clinical study within 30 days prior to day-of-surgery or plans to participate in another clinical study while concurrently enrolled in this study.
15. Subject has a history of conditions which might be specifically contraindicated or require caution to be used during the administration of any drug in the study.
16. Subject has any other medical, psychiatric and/or social reason for exclusion as determined by the investigator.
17. Subject has a positive test result for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids [including medical use of marijuana], cocaine, methamphetamine, methadone, or methylenedioxy-methamphetamine) at Screening. Subjects with a positive test result for prescribed drugs may be included in the study at the discretion of the investigator. Subjects with a positive test result for cannabinoids with a prescription for medical marijuana will be excluded from the study, subjects with a prescription for dronabinol (∆-9-tetrahydrocannabinol) may be included at the discretion of the investigator.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2016-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Mallinckrodt
Locations (2):
- United States (2):
  - Pensacola Research Consultants, Pensacola, Florida
  - The Ohio State University, Wexner Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Acetaminophen/Morphine: IV acetaminophen 1000 mg every 6 hours over 18 hours
  IV acetaminophen
  Morphine: Patient controlled analgesia
- Oral Acetaminophen/Morphine: Oral acetaminophen two 500 mg tablets every 6 hours over 18 hours
  Oral acetaminophen
  Morphine: Patient controlled analgesia
Period: Overall Study
Arm/Group | IV Acetaminophen/Morphine | Oral Acetaminophen/Morphine
Started | 0 | 1
Per Protocol Analysis Set | 0 | 0
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Per Protocol Analysis Set - The single participant enrolled was in violation of the protocol, leading to unreliable or uninterpretable data.
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen/Morphine | Oral Acetaminophen/Morphine | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity on a Numerical Pain Scale (NPS) for 18 Hours
Description: Participants rate intensity of their pain on a Numerical Pain Scale (NPS) from 0-10, wherein 0=no pain (better) and 10=most intense pain (worse). The highest possible score is 10.
Time Frame: 18 hours
Population: as for baseline characteristics
Arm/Group | IV Acetaminophen/Morphine | Oral Acetaminophen/Morphine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 days
Description: Number of participants at risk for All-Cause Mortality, Serious Adverse Events (SAEs) and Non-serious Adverse Events (AEs) are all 0 for the intravenous acetaminophen arm because no participants were enrolled into that arm. All non-serious AEs are reported for the single subject enrolled into the oral acetaminophen arm (including opioid AEs).
Arm/Group | IV Acetaminophen/Morphine | Oral Acetaminophen/Morphine
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Acetaminophen/Morphine (N=0) | Oral Acetaminophen/Morphine (N=1)
Acute blood loss anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diffuse bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Intermittent thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Intermittent leucocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Persistent sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Postoperative pain (General disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stress hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1)
Suspicion of adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small number of participants analyzed.

The single participant enrolled was in violation of the protocol, leading to unreliable or uninterpretable data.

All AEs were listed, but not related to the study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes